CLINICAL TRIAL: NCT06252207
Title: Desflurane Versus Isoflurane for Speeding Postanesthetic Recovery and Hospital Discharge: a Cluster Randomized Crossover Trial
Brief Title: Desflurane Versus Isoflurane for Speeding Postanesthetic Recovery and Hospital Discharge
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The Cleveland Clinic (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Other
Other Study IDs: 23-1049
Record Dates: First submitted 2024-01-22; First posted 2024-02-09 (Actual); Last update posted 2025-08-11 (Actual); Status verified 2025-08

CONDITIONS: Surgery
MeSH Terms: interventions — Desflurane; Isoflurane

STUDY DESIGN:
Intervention Model Description: Randomized cluster cross-over trial
Who Masked: Participant
Masking Description: Patients will not be told which type of volatile anesthetic they received.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Desflurane (Experimental): General anesthesia with desflurane.
  Interventions: Drug: Desflurane
- Isoflurane (Experimental): General anesthesia with isoflurane.
  Interventions: Drug: Isoflurane

INTERVENTIONS:
Drug: Desflurane — General anesthesia with desflurlane
  Arms: Desflurane
Drug: Isoflurane — General anesthesia with isoflurane
  Arms: Isoflurane

SUMMARY:
The investigators thus propose a comparative effectiveness quality improvement project to evaluate the feasibility of switching from near-exclusive use of isoflurane in adult general surgical patients to Desflurane.

DETAILED DESCRIPTION:
The three available volatile anesthetics appear to be comparably safe. However, higher solubility slows emergence from isoflurane and sevoflurane compared to Desflurane. Even a few minutes delay in emergence from anesthesia has financial implications since institutional costs of operating room time can easily be $30 per minute. Postoperative care is also expensive. Furthermore, in busy hospitals such as the Cleveland Clinic, inadequate recovery throughput frequently delays surgery.

The investigators thus propose a comparative effectiveness quality improvement project to evaluate the feasibility of switching from near-exclusive use of isoflurane in adult general surgical patients to Desflurane. (The investigators will exclude children because there are compelling clinical reasons to use sevoflurane in pediatric patients.) The proposed comparison is between isoflurane (our current routine) and Desflurane which is no longer used at the Clinic because of price concerns - a decision that that did not consider down-stream effects, including prolonged emergence and recovery.

ELIGIBILITY:
Inclusion Criteria:

* Adults having general anesthesia in the G operating room suite at the Cleveland Clinic Main Campus.

Exclusion Criteria:

* Operations lasting <1.5 hours.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2619 (Estimated)
Dates: Start 2023-12-08 (Actual); Primary Completion 2026-03-01 (Estimated); Study Completion 2026-12-01 (Estimated)

PRIMARY OUTCOMES:
Duration of post-anesthesia care unit recovery | 1 hour
  Time from entry to the post-anesthesia to discharge from unit.

SECONDARY OUTCOMES:
Duration of anesthetic emergence | 1 hour
  Time from a MAC fraction of 0.3 (presumably shortly after volatile anesthesia is discontinued) and extubation.
Cost of post-anesthesia care unit. | 2 hours
  Cost of post-anesthesia unit care. To be estimated only if there is a substantial difference between the groups.
Delirium | 5 days
  Incidence of postoperative delirium.

CONTACTS AND LOCATIONS:
Overall Officials: Allen Keebler, D.O., Principal Investigator — The Cleveland Clinic
Locations (1):
- Cleveland Clinic, Cleveland, Ohio, United States

IPD SHARING:
Plan to Share IPD: No